CLINICAL TRIAL: NCT02687893
Title: A Randomized, Three-way, Cross-over Study to Assess the Impact of Nocturnal Hypoglycemia on Sleep in Patients With Type 1 Diabetes
Brief Title: Effect of Hypoglycemia on Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Peter G. Jacobs, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15228
Record Dates: First submitted 2016-01-25; First posted 2016-02-22 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Hypoglycemia
Keywords: Sleep; Exercise
MeSH Terms: conditions — Hypoglycemia; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aerobic Exercise Week (Experimental): Subjects will complete 45 minutes of aerobic exercise twice during a 7 day period. Exercise will be graded based on the participant's relative capacity determined at the screening visit. Each exercise session will be followed by 60 minutes of monitored resting recovery.
  Interventions: Behavioral: Aerobic Exercise
- Resistance Exercise Week (Experimental): Subjects will complete 45 minutes of anaerobic exercise twice during a 7 day period. Each exercise session will be followed by 60 minutes of monitored resting recovery.
  Interventions: Behavioral: Resistance Exercise
- No Exercise Week (No Intervention): Subjects will perform no exercise during this week.

INTERVENTIONS:
Behavioral: Aerobic Exercise — Subjects will exercise on a treadmill for 45 minutes twice during the intervention week. Subjects will exercise at a fixed intensity level to a target heart rate (±10%) based on the heart rate achieved at 60% of their VO2max determined at screening. The speed and grade of the treadmill will be adjusted by trained research personnel with a goal of keeping participants within their target heart rate range for the entire 45 minutes.
  Arms: Aerobic Exercise Week
Behavioral: Resistance Exercise — Subjects will participate in resistance exercises for 45 minutes twice during the intervention week. Subjects will perform multiple-joint exercises with slow to moderate lifting velocity, for 1-3 sets per exercise at a weight that can be lifted for 8-12 repetitions (~60-80% of 1-repetition max). The exercises may include leg press, bench press, leg extension, leg flexion and seated row. Subjects will perform the exercises through the full range of motion. Between each set of repetitions, there would be a 2 minute rest period. The duration of the exercise testing would be approximately 45 minutes.
  Arms: Resistance Exercise Week

SUMMARY:
Growing evidence provided by many observational studies has established a strong link between decreased sleep duration and poor glucoregulation. Sleep deprivation and poor sleep quality induce insulin resistance and decrease glucose tolerance in healthy individuals. However, the influence of poor sleep quality on glycemic control of patients with Type 1 diabetes mellitus (T1DM) is unknown. Persistent sleep deprivation among patients with T1DM has been reported, and this sleep loss can be attributed in part to nocturnal hypoglycemia. Nocturnal iatrogenic hypoglycemia is a limitation of current intensive insulin therapies. Although severe hypoglycemia is associated with adverse events such as seizures and death, less severe nocturnal hypoglycemia has been linked to broad range of adverse consequences, both acutely and long term. Hypoglycemia stimulates the sympathetic nervous system as a stress response, leading to the stimulation of the hypothalamic-pituitary-adrenal axis (HPA). This results in a counter regulatory hormone cascade, which elicits an excessive cortisol secretion, which is known to cause sleep disturbance and could impair glucose homeostasis after the hypoglycemic event. The hyperinsulinemia in T1DM patients promotes HPA hyperactivity as well, which is also associated with impaired sleep quality by leading to sleep fragmentation, decreased slow wave sleep and shortened sleep duration. Sleep disturbances due to nocturnal hypoglycemia can exacerbate HPA axis dysfunction, adversely affecting the sleep-wake cycle.

The goal of the study is to understand the impact of nocturnal hypoglycemia on sleep.

DETAILED DESCRIPTION:
The study duration is 4 weeks long, during which subjects will undergo a 1 week run-in period followed by 3 randomized weeks of observational study. During the 1 week run-in period, subjects will familiarize themselves with the CGM and the other data collection procedures. Following the run-in week, the subject will be randomized to a specific order of observation weeks. The three observation weeks are a resistance training week, an aerobic exercise week and a control week with no explicit exercise. During the observation weeks, there will be 4 interventions planned, two during both the aerobic exercise and the resistance training week. See Schematic below for details. During both the aerobic exercise week intervention visits, subjects will exercise for ~45 minutes on a treadmill and during the resistance training week, subjects will perform strength training exercises for 1-3 sets per exercise at a weight that can be lifted for 8-12 repetitions (~60-80% of 1-repetition max). The duration of the resistance training period is expected to be ~45min. Subjects will continue to perform daily activities during each of the weeks.

During each week, the subject will wear one subcutaneous DexcomTM G4 or DexcomTM G4 Share continuous glucose monitoring (CGM) system, one activity monitor- ActiGraph wGT3X-BT or ActiGraph GT9X, one insulin pump (subject's own pump) and one Samsung Galaxy S4 phone loaded with two applications- meal memory and moves. The CGM system will provide sensed glucose data every 5 minutes. The CGM data will be blinded to the patient to prevent any abrupt changes in behavior. The accuracy of the sensed data will be obtained by reference measurements of capillary blood glucose. The activity monitor will be secured on the dominant wrist and uses an accelerometer to collect movement data at a high frequency (80Hz). The activity monitor measures both motion and ambient light, this data would be used to determine the various sleep quality measures. The subject's insulin dosage information from the pump will be downloaded for data analysis purposes. The subject's daily meal intake (photographic log and note diary) and daily movement pattern information will be downloaded from the phone. During the 4 exercise intervention visits, subject's heart rate, accelerometry information from the torso and oxygen consumption measured breath by breath may be collected for data analysis purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 1 diabetes mellitus for at least 1 year.
2. Male or female subjects 21 to 45 years of age.
3. Physically active on a regular basis, i.e. at least 3 days of physical activity per week.
4. Physically willing and able to perform 45 min of exercise (as determined by the investigator after reviewing the subjects activity level)
5. Current use of an insulin pump.
6. Willingness to follow all study procedures, including attending all clinic visits.
7. Willingness to sign informed consent and HIPAA documents.

Exclusion Criteria:

1. Female of childbearing potential who is pregnant or intending to become pregnant or breast-feeding, or is not using adequate contraceptive methods. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an intrauterine device (IUD), the double barrier method (the woman uses a diaphragm and spermicide and the man uses a condom), or abstinence.
2. Any cardiovascular disease, defined as a clinically significant EKG abnormality at the time of screening or any history of: stroke, heart failure, myocardial infarction, angina pectoris, or coronary arterial bypass graft or angioplasty. Diagnosis of 2nd or 3rd degree heart block or any non-physiological arrhythmia judged by the investigator to be exclusionary.
3. Renal insufficiency (GFR < 60 ml/min, using the MDRD equation as report by the OHSU laboratory).
4. Impaired liver function, defined as AST or ALT ≥2.5 times upper limit of normal, according to OHSU laboratory reference ranges.
5. Hematocrit of less than or equal to 34%.
6. History of severe hypoglycemia during the past 12 months prior to screening visit or hypoglycemia unawareness as judged by the investigator.
7. Adrenal insufficiency.
8. Any active infection.
9. Known or suspected abuse of alcohol, narcotics, or illicit drugs (except marijuana use).
10. Seizure disorder.
11. Active foot ulceration.
12. Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication.
13. Major surgical operation within 30 days prior to screening.
14. Use of an investigational drug within 30 days prior to screening.
15. Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
16. Bleeding disorder, treatment with warfarin, or platelet count below 50,000.
17. Insulin resistance requiring more than 200 units per day.
18. Need for uninterrupted treatment with acetaminophen.
19. Current administration of oral or parenteral corticosteroids.
20. Any life threatening disease, including malignant neoplasms and medical history of malignant neoplasms within the past 5 years prior to screening (except basal and squamous cell skin cancer).
21. C peptide level of ≥0.5 ng/ml
22. Any concurrent illness, other than diabetes, that is not controlled by a stable therapeutic regimen.
23. Beta blockers or non-dihydropyridine calcium channel blockers.
24. A positive response to any of the questions from the Physical Activity Readiness Questionnaire.
25. Any chest discomfort with physical activity, including pain or pressure, or other types of discomfort.
26. Any clinically significant disease or disorder which in the opinion of the Investigator may jeopardize the subject's safety or compliance with the protocol.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02; Primary Completion 2016-09 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Mean duration of time with sensed glucose less than 70 mg/dl post-exercise | 16 hours
  The mean duration of time in hypoglycemia in minutes (defined as sensor glucose less than 70 mg/dl) will be calculated using sensor glucose data acquired by the Dexcom G4 for 16 hours after the beginning of exercise.

SECONDARY OUTCOMES:
Mean duration with sensed glucose between 70 - 180 mg/dl post-exercise | 16 hours
  The mean duration of time in euglycemia in minutes (defined as sensor glucose between 70-180 mg/dl) will be calculated using sensor glucose data acquired by the Dexcom G4 for 16 hours after the beginning of exercise.
Mean duration with capillary blood glucose between 70 - 180 mg/dl | 4 weeks
  The mean duration of time in euglycemia in minutes (defined as capillary blood glucose between 70-180 mg/dl) will be calculated using blood glucose data acquired by the Contour Next blood glucose (BG meter.
Mean wake up after sleep onset duration post-exercise | 16 hours
  Using data acquired from an Actigraph activity monitor, mean duration of time in minutes of wake after sleep onset for the 16 hours after the beginning of exercise.
Mean amplitude of glucose excursions | 4 weeks
  The mean amplitude of glucose excursions will be calculated using sensor glucose data acquired by the Dexcom G4.
Mean duration of total sleep time | 4 weeks
  Using data acquired from an Actigraph activity monitor, mean duration of time in minutes that subject is asleep.
Mean time subject in bed | 4 weeks
  Using data acquired from an Actigraph activity monitor, mean duration of time in minutes that subject is in bed.
Mean time for sleep onset | 4 weeks
  Using data acquired from an Actigraph activity monitor, mean duration of time in minutes associated with the first epoch of the first 10 minute period of immobility starting from lights out time.
Mean time of sleep efficiency | 4 weeks
  Using data acquired from an Actigraph activity monitor, a ratio of total sleep time to assumed sleep time multiplied by 100.
Mean number of wake bouts | 4 weeks
  Using data acquired from an Actigraph activity monitor, mean of continuous blocks of length greater than or equal to 1 epoch in which each epoch is scored as wake in the assumed sleep period.
Mean wake bout time | 4 weeks
  Using data acquired from an Actigraph activity monitor, mean time in minutes of wake after sleep onset divided by the number of wake bouts.
Mean number of sleep bouts | 4 weeks
  Using data acquired from an Actigraph activity monitor, mean of continuous blocks of length greater than or equal to 1 epoch in which each epoch is scored as sleep in the assumed sleep period.
Mean sleep bout time | 4 weeks
  Using data acquired from an Actigraph activity monitor, mean time in minutes of total sleep time divided by the number of sleep bouts.
Mean number of carbohydrate treatments to treat hypoglycemia | 4 weeks
  Number of rescue carbohydrate treatments administered by the subject through study completion.
Mean daily carbohydrate intake | 4 weeks
  Measuring the number of grams of carbohydrates consumed by the subjects through study completion.
Mean daily insulin intake | 4 weeks
  Measuring the number of units of insulin administered to the subject by his/her insulin pump through study completion.
Mean of total duration of activity by the subject | 4 weeks
  Using data acquired from an Actigraph activity monitor, mean duration of time in minutes of activity by the subject through study completion.
Mean duration of time with sensed glucose < 50 mg/dl | 4 weeks
  The mean duration of time in hypoglycemia in minutes (defined as sensor glucose below 50 mg/dl) will be calculated using sensor glucose data acquired by the Dexcom G4.
Mean duration of time with capillary blood glucose < 50 mg/dl | 4 weeks
  The mean duration of time in hypoglycemia in minutes (defined as capillary blood glucose below 50 mg/dl) will be calculated using capillary blood glucose data acquired by the Contour Next BG meter.
Mean duration of time with capillary blood glucose < 70 mg/dl | 4 weeks
  The mean duration of time in hypoglycemia in minutes (defined as capillary blood glucose below 70 mg/dl) will be calculated using capillary blood glucose data acquired by the Contour Next BG meter.
Mean duration of time with sensed glucose > 180 mg/dl | 4 weeks
  The mean duration of time in hyperglycemia in minutes (defined as sensor glucose greater than 180 mg/dl) will be calculated using sensor glucose data acquired by the Dexcom G4.
Mean duration of time with capillary blood glucose > 180 mg/dl | 4 weeks
  The mean duration of time in hyperglycemia in minutes (defined as blood glucose greater than 180 mg/dl) will be calculated using glucose data acquired by the Contour Next BG meter.

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Jacobs, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No